CLINICAL TRIAL: NCT02659202
Title: Spinal Cord Stimulation to Inhibit Afferent Feedback During Exercise in Heart Failure
Brief Title: Spinal Stimulation During Exercise in Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to continue the study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Johnson, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-002521
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Exercise; Heart Failure; Blood Pressure
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Precision Spinal Cord Stimulator System (Experimental): Intervention:the precision system will consist of a pulse generator that will not be implanted, temporary percutaneous leads lead extensions, each packaged as a separate kit.
  Interventions: Device: Precision Spinal Cord Stimulator System

INTERVENTIONS:
Device: Precision Spinal Cord Stimulator System — The precision system will consist of a pulse generator that will not be implanted, temporary percutaneous leads, surgical paddle leads and lead extensions, each packaged as a separate kit.

SUMMARY:
The purpose of this proposal is to determine whether epidural spinal cord stimulation can modulate cardiovascular control during exercise in Heart Failure patients.

DETAILED DESCRIPTION:
Forty Heart Failure (>18 yrs. of age) will be recruited. The study will include a total of 2 visits. All experiments will take place at the Mayo Clinic; at the outpatient radiology for MRI screening, the Charlton Clinical Research Unit (CRU) for surgical suite for spinal cord stimulation placement and the Saint Mary's Hospital Clinical Research Unit for clinical exercise laboratory for the exercise protocol and overnight stay.

Study visit 1 will include eligibility screening, consenting process, completion of a health questionnaire and performance of a peak oxygen consumption (VO2) test. Additionally, subjects will undergo a screening lumbar MRI to ensure that there are no anatomical anomalies in or around the epidural area consistent with standard clinical practice for epidural stimulator lead placement associated with chronic pain syndromes.

Study visit 2 will include an overnight stay in the Saint Mary's Hospital Clinical Research Unit. Patients will check in to the CRU in the morning of day 1, visit 2. Prior to placement of stimulating electrodes an international normalized ratio (INR) will be checked to ensure safe clotting. An anesthesiologist will place the electrodes in the lumbar/thoracic epidural space in a manner that is standard for the clinical placement of temporary electrodes in humans. The participants will then transfer to the clinical exercise laboratory to start the exercise protocol. Participants will rest 15 minutes prior to starting exercise. Exercise will take place on a vertical bike where they will perform a submaximal cycling exercise at 30% of peak work for 29 minutes. Thigh cuffs will be placed on thigh bilaterally and inflated intermittently to pressures of 80m mmHg. After the testing is complete, participants will return to their room in the Clinical Research Unit for the rest of the day and sty over night.

On day two of visit two, participants will repeat the testing from day one with new randomization to determine reliability of testing performed on day one. After the exercise on day two of visit two, the spinal cord stimulator leads and radial arterial catheter will be removed.

ELIGIBILITY:
Inclusion Criteria, includes:

* Heart Failure patients with reduced ejection fraction:
* History of ischemic or idiopathic dilated cardiomyopathy (duration > 1yr.) stable for > 3mo and New York Heart Association Class I-III
* Not pacemaker dependent
* Body Mass Index ≤35
* Ejection Fraction < 40%
* Current nonsmokers with < 15 pack year history
* Able to exercise

Exclusion Criteria includes:

* History of cardiopulmonary disorders and dangerous arrhythmias
* Pregnant women
* Taking prescribed opioid medications or have had a fusion or laminectomy at L3 or above
* Patients with a recent drug-eluding stent
* History of spinal stenosis, lumbar radiculopathy, or peripheral neuropathy
* Must not currently be taking blood thinners or anticoagulant medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Johnson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precision Spinal Cord Stimulator System
Started | 7
Completed | 3
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Precision Spinal Cord Stimulator System
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Description: This will allow for continuous real-time intra-arterial measurement of beat-to-beat blood pressure.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Precision Spinal Cord Stimulator System
Number analyzed (Participants) | 3
mmHg | 82.3 (10.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from enrollment through the end of the final visit, for approximately 1 month.
Arm/Group | Precision Spinal Cord Stimulator System
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulator System (N=7)
Paresthesia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT02659202/Prot_SAP_000.pdf